CLINICAL TRIAL: NCT01606618
Title: Analysis of Psychosocial Determinants of Observance of Monitoring Neuro-urological in Spina-bifida Adult Patients and in Spinal Cord Injury Patients: a Prospective, Comparative, Multicenter With Parallel Groups Study
Brief Title: Self-esteem and Neuro-urological Follow-up in Patients With Spina Bifida or Spinal Cord Injury
Acronym: ESTIME
Status: Terminated | Type: Observational
Why Stopped: Sponsor and investigator's decision
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: B110797-30
Record Dates: First submitted 2012-05-16; First posted 2012-05-28 (Estimated); Last update posted 2021-04-15 (Actual); Status verified 2021-04

CONDITIONS: Spina Bifida Aperta; Acquired Traumatic Spinal Cord Injury
Keywords: Self-esteem; Spina Bifida; Spinal cord injury
MeSH Terms: conditions — Spina Bifida Cystica; Spinal Dysraphism; Spinal Cord Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Spina bifida aperta
- Acquired traumatic spinal cord injury

SUMMARY:
With improved life expectancy over the last fifty years, spina bifida has become a disease of the adult. One of the major stakes for these patients is the preservation of a regular follow-up of uro-nephrologicals risk factors and of a respect for the rules of self management of their neurological bladder.

The main objective of this study is to highlight a difference in the level of global self-esteem among a population of adult patients with spina bifida and a population of adult patients with traumatic spinal cord injury gained the same level of neurological.

DETAILED DESCRIPTION:
With improved life expectancy over the last fifty years, spina bifida has become a disease of the adult. The risk of developing a terminal renal insufficiency is eight times higher than the risk in the general population and twice as important as in acquired spinal cord injury. This risk continues to evolve with advancing age.

One of the major stakes for these patients is the preservation of a regular follow-up of uro-nephrologicals risk factors and of a respect for the rules of self management of their neurological bladder. However, some studies report that nearly two thirds of these patients are not monitored at regular neuro-urological in the adulthood. Different psychosocial determinants were analyzed as potential markers of the impact of chronic diseases from childhood to adulthood and could account for the disparity of follow-up and access to healthcare. Among these, the self-esteem is a psychological dimension of analysis particularly relevant within the framework of chronic states inherited from the childhood.

The investigators formulate the hypothesis that global self-esteem and lower perceived self-efficacy may be a causal predictive factor of a reduced access to the continence and a lower compliance monitoring in adult patients with a spina bifida.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a spina bifida aperta or an acquired traumatic spinal cord injury dating more than two years, the level of injury being below D12 and higher S1 (Score ASIA A).
* Age between 18 and 60
* Knowing how to read, write, count
* Having given their free, informed and in writing consent (an information is also given to the reliable person when it exists)
* Affiliated to the National Health Service

Exclusion Criteria:

* Psychiatric history requiring an hospitalization in a specialized unit during more than two months
* Score MMS lower than 27 ( GRECO version)
* Serious associated pathology or associated pathology which could interfer with the management of vesico-sphincteral disorders
* Neurosurgery, dating from less than one year
* Symptoms of dysfunction of ventricular bypass valve at the time of inclusion
* Clinical epileptic attack within six months prior to inclusion
* Pregnancy or breastfeeding
* Simultaneous inclusion in an another therapeutic protocol or period of exclusion from an another protocol
* Traumatic spinal cord injury acquired before age 16

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patient seen in university hospitals or in rehabilitation clinic
Sampling Method: Non-Probability Sample
Enrollment: 111 (Actual)
Dates: Start 2012-03-12 (Actual); Primary Completion 2017-09-11 (Actual); Study Completion 2017-09-11 (Actual)

PRIMARY OUTCOMES:
Measure of the global self-esteem by the Rosenberg scale (RSES) | At day 0
  Score range : 10 - 40. High scores indicate hight self esteem.

SECONDARY OUTCOMES:
Evaluation of depression and anxiety by Hamilton's scale (HAD) | At day 0, at month 6
  Score range : 0 - 21. High scores indicate a hight level of symptoms.
Neuropsychological evaluation (WAIS-III battery composite GREFEX, CVLT) | At day 0
  Battery of test exploring executives functions. High scores indicate high level of executive functions.
Rating Scale vesico-sphincter and anorectal function (ISCOS) | At day 0, at month 6
  High scores indicate high vesico-sphincter and anorectal dysfunction
Evaluation scale for the achievement of self catheterizing | At day 0, at month 6
  14 binary items
Scale functional mobility and transfers (SCIM III) | At day 0
  The SCIM is a disability scale in order to describe patients' ability to accomplish activities of daily living and to make functional assessments of this population more sensitive to changes.
  SCIM-III is comprised of 19 items in 3 subscales, which are:
  (i) self-care (sub-score 0-20); (ii) respiration and sphincter management (sub-score 0-40); (iii) mobility (sub-score 0-40). The mobility subscale is further sub-divided to assess mobility "in room and toilet" and for "indoors and outdoors, on an even surface".
  The total score ranges from 0 to 100.
Measure of the global self-esteem by the Rosenberg scale (RSES) | At month 6
  Score range : 10 - 40. High scores indicate hight self esteem.
Observance of the appointment | At month 6
Observance of holding of the mictionnel catalog | At month 6
Measure of auto-efficiency experienced scale for Medullary Injured (MSES) | At Day 0
  * 16 items ranging from 1 to 7
  * Range 16 - 112
  * High scores correspond to low level of percieved auto-efficiency

CONTACTS AND LOCATIONS:
Overall Officials: Jacques Kerdraon, MD, Principal Investigator — CHU Rennes; Reymann Jean Michel, PhD, Study Chair — Rennes University Hospital
Locations (16):
- France (16):
  - CHU de Besançon, Besançon
  - Clinique Saint Augustin, Bordeaux
  - CHU de Lille, Lille
  - Urologie CH Lyon Sud et Hôpital Henry Gabrielle, Lyon
  - APHM - Hôpital de la Conception Service de chirurgie urologique et transplantation rénale, Marseille
  - MPR neurologique CHU de Nantes, Nantes
  - APHP Raymond Poincaré, Paris
  - APHP Rothschild, Paris
  - Neuro-urologie et explorations périnéales, APHP Tenon, Paris
  - Centre Mutualiste de Rééducation et de Réadaptation Fonctionnelles de KERPAPE, Ploemeur
  - CHU de Rennes CR Spina bifida, Rennes
  - Hôpital Pontchaillou - CHU de Rennes, Rennes
  - MPR St Hélier, Rennes
  - Urologie, CHU de Rouen, Rouen
  - MPR CHU Rangueuil, Toulouse
  - Urologie CHU Rangueuil Toulouse, Toulouse